CLINICAL TRIAL: NCT01649453
Title: A Prospective Study of Clinical Outcomes for the Pathwork® Tissue of Origin Test
Brief Title: A Prospective Study of Clinical Outcomes for the Pathwork Tissue of Origin Test
Status: Terminated | Type: Observational
Why Stopped: Terminated by sponsor.
Sponsor: Cedar Associates LLC (Other)
Collaborators: Pathwork Diagnostics (Unknown)
Responsible Party: Principal Investigator, John Hornberger, MD MS, CEO, President, Cedar Associates LLC
Other Study IDs: 10043P
Record Dates: First submitted 2012-07-23; First posted 2012-07-25 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Neoplasm Metastasis
Keywords: Neoplasms; Neoplasm Metastasis; Neoplastic Processes; Pathologic Processes
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms; Neoplastic Processes; Pathologic Processes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue biopsy specimen.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cancer of uncertain primary
  Interventions: Device: Pathwork® Tissue of Origin Test

INTERVENTIONS:
Device: Pathwork® Tissue of Origin Test
  Other Names: Gene expression profile tissue of origin test

SUMMARY:
The study prospectively assesses the change in cancer-specific clinical decisions and outcomes before and after physicians received results from the Pathwork® Tissue of Origin (TOO) Test for patients whose primary site of cancer origin is uncertain.

ELIGIBILITY:
Inclusion Criteria:

* their physician ordered or intends to order a Pathwork® TOO Test between May 2012 and December 2013
* the patient is ≥ 18 years of age
* the patient has given informed consent (online or verbal)
* the patient is able to understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community and academic clinics
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: John Hornberger, MD MS, Principal Investigator — Cedar Associates LLC
Locations (1):
- Cedar Associates LLC, Menlo Park, California, United States